CLINICAL TRIAL: NCT01831609
Title: Biomarker Analysis of Solid Cancers Such as Gastrointestinal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, Assistant Professor, Samsung Medical Center
Other Study IDs: 2011-07-089-013
Record Dates: First submitted 2013-04-07; First posted 2013-04-15 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Sarcoma
Keywords: Gastrointestinal; Genitourinary; Rare Cancer
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pleural fluid, ascites, fine needle aspirations, other body fluids (i.e. CSFs)prospectively. Primary cultures, Xenografts.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To prospectively collect ascites, pleural fluid, circulating tumor cells and derived primary cultures from metastatic cancer patients. The specimens will be analyzed using DNA/RNA/proteomic approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed gastrointestinal, genitourinary, sarcoma, rare cancer
2. Written informed consent
3. body fluid derived from cancer, available for drainage and collection

Exclusion Criteria:

* patients who do not give informed consent form for research use of biomaterials/biospecimens

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Patients with histologically confirmed gastrointestinal, genitourinary, sarcoma, rare cancer
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-08-31 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Biomarker analyses to predict treatment response in metastatic cancer | 3 year
  Using patient derived tumor cells, predictive biomarker analyses (DNA, RNA protein levels etc) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jeeyun Lee, professor, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea